CLINICAL TRIAL: NCT02927808
Title: Motivational Interviewing to Support LDL-C Therapeutic Goals and Lipid-Lowering Therapy Compliance in Patients With Acute Coronary Syndromes: a Prospective Randomized Clinical Study
Acronym: IDEAL-LDL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AHEPA University Hospital (Other)
Responsible Party: Principal Investigator, Leonidas Lillis, MD, Clinical Research Associate, AHEPA University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22904/25.5.2016
Record Dates: First submitted 2016-10-06; First posted 2016-10-07 (Estimated); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Acute Coronary Syndrome
Keywords: Motivational Interviewing; LDL-C; LDL target; Medication adherence
MeSH Terms: conditions — Acute Coronary Syndrome; Medication Adherence | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group - Motivational Interview (Experimental): Patients assigned to the intervention group will be given a leaflet entitled "Information leaflet about LDL Cholesterol" that will educate them about the risks of high LDL-C and the importance of adherence to lipid-lowering medication. Patients assigned to the intervention group will be contacted via telephone for a pre-specified interview (motivational interview again stressing the importance of adherence to lipid-lowering medication) at 1 month and 6 months after discharge, and for an in-person interview plus lipid profiling at 1 year after discharge.
  Interventions: Behavioral: Motivational Interview
- Control group (No Intervention): Patients assigned to the control group will be contacted for a pre-specified in-person interview plus lipid profiling at 1 year after discharge.

INTERVENTIONS:
Behavioral: Motivational Interview — Informational leaflet about the risks of high LDL-C and the importance of adherence to lipid-lowering medication in patients with coronary artery disease. Follow-up motivational interviewing at 1 and 6 months after discharge.
  Arms: Intervention group - Motivational Interview

SUMMARY:
This study will investigate the impact of motivational interviewing in achieving low-density lipoprotein cholesterol therapeutic targets in patients with acute coronary syndromes.

DETAILED DESCRIPTION:
To determine whether a strategy of enhanced information about the risks of high plasma low-density lipoprotein cholesterol (LDL-C) and the importance of lipid-lowering medication together with close follow-up and motivational interviewing is superior than usual care in achieving LDL-C therapeutic targets, as set by current practice guidelines (LDL-C <70 mg/dL or >50% reduction from baseline LDL-C) in patients with acute coronary syndromes.

ELIGIBILITY:
Inclusion Criteria:

* Subject hospitalized for acute coronary syndrome (STEMI, NTEMI or unstable angina)
* Subject currently on lipid-lowering therapy or prescribed lipid-lowering therapy at hospital discharge (statins and/or other agents)
* Subject who is 18 years or older
* Subject or legally authorized representative who is willing and capable of providing informed consent, participating in all associated study activities

Exclusion Criteria:

* Subject unable to communicate via telephone for study interviewing
* Subject with contraindication to statin therapy
* Subject with any medical disorder that would interfere with completion or evaluation of clinical study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Achievement of low-density lipoprotein cholesterol therapeutic goal, as specified by current practice guidelines (LDL-C <70 mg/dL or >50% reduction from baseline LDL-C) | 12 months after discharge from hospital

SECONDARY OUTCOMES:
Overall adherence to lipid-lowering regimen, reported as both a continuous and a binary outcome, by using the 4-item Morisky Medication-Taking Adherence Scale | 12 months after discharge from hospital

CONTACTS AND LOCATIONS:
Locations (1):
- AHEPA University Hospital, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kourti O, Konstantas O, Farmakis ITau, Zafeiropoulos S, Psarakis G, Vrana E, Baroutidou A, Graidis S, Touriki AV, Tsolakidis C, Spyridaki K, Psathas T, Daniilidou A, Karvounis H, Giannakoulas G. Potent P2Y12 inhibitors versus clopidogrel to predict adherence to antiplatelet therapy after an acute coronary syndrome: insights from IDEAL-LDL. Rev Cardiovasc Med. 2022 Mar 3;23(3):81. doi: 10.31083/j.rcm2303081. PMID 35345248
- [Derived] Zafeiropoulos S, Farmakis I, Kartas A, Arvanitaki A, Pagiantza A, Boulmpou A, Tampaki A, Kosmidis D, Nevras V, Markidis E, Papadimitriou I, Vlachou A, Arvanitakis K, Miyara SJ, Ziakas A, Molmenti EP, Kassimis G, Zanos S, Karvounis H, Giannakoulas G. Reinforcing adherence to lipid-lowering therapy after an acute coronary syndrome: A pragmatic randomized controlled trial. Atherosclerosis. 2021 Apr;323:37-43. doi: 10.1016/j.atherosclerosis.2021.03.013. Epub 2021 Mar 17. PMID 33780749